CLINICAL TRIAL: NCT03817112
Title: The Effect of Continuous Propofol Versus Dexmedetomidine Infusion on Regional Cerebral Tissue Oxygen Saturation During Cardiopulmonary Bypass
Brief Title: Effect of Dexmedetomidine and Propofol on Regional Cerebral Tissue Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Clinical professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASCSH86/17
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Regional Cerebral Tissue Oxygen Saturation
Keywords: cerebral oxygen saturation; cardiopulmonary bypass; dexmedetomidine; propofol
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Infusion of dexmedetomidine
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.1 MG/ML
- Propofol (Active Comparator): Propofol infusion
  Interventions: Drug: Propofol 10 MG/ML

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride 0.1 MG/ML — Dexmedetomidine Hydrochloride 0.1 MG/ML infusion at 0.2-0.7 mcg/kg/min
  Arms: Dexmedetomidine
Drug: Propofol 10 MG/ML — Propofol 10 MG/ML infusion at 0.3 -4 mg/kg/h
  Arms: Propofol

SUMMARY:
50 patients divided into 2 groups

.Group I Dexmedetomidine infusion. Group II with Propofol infusion

DETAILED DESCRIPTION:
: 50 patients anticipated for open heart surgeries were encompassed in the study. Patients were divided into 2 groups, group P (receiving propofol) and group D (receiving dexmedetomidine) during CPB. Both groups were studied for variations in right and left rScO2 as well as postoperative cognitive dysfunction using the Mini Mental State Examination Score (MMSE) test.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing valve surgeries
* Patients undergoing on pump coronary artery bypass grafting surgeries

Exclusion Criteria:

* emergency cases, patients with cervical spine pathology (cervical stenosis, cervical disc herniation, carotid stenosis), patients with cerebral pathology (cerebral strokes, ischemic attacks), patients with Mini Mental State Examination Score (MMSE) of 23 or less, complicated cases with prolongation of the cardiopulmonary bypass period, patients needing moderate hypothermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
cognitive function assessment | 24 hours postoperative
  Mini Mental State Examination Score (MMSE) test to assess orientation to time and place with ability to speak, think and draw. with highest ability 32 and lowest o

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Cardiothoracic hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No